CLINICAL TRIAL: NCT00793767
Title: Insulin Resistance and Substrate Metabolism After Acute EPO Administration in Healthy Young Men
Brief Title: Insulin Resistance and Substrate Metabolism After Acute Erythropoietin (EPO) Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Phd. student, Britt Christensen, Afdeling M, Århus sygehus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: M-20080016
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Insulin Sensitivity
Keywords: Erythropoietin; human muscle tissue; insulin sensitivity; substrate metabolism
MeSH Terms: conditions — Insulin Resistance | interventions — Erythropoietin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo (saline)
- Erythropoietin (Experimental): acute administration of erythropoietin
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: erythropoietin — bolus of 400 IU/kg
  Arms: Erythropoietin
Drug: placebo (saline) — i.v
  Arms: placebo

SUMMARY:
Recently EPO receptors have been found in human muscle tissue, but what is still not known is the physiological role of these receptors. In this study the researchers want to investigate if there is any effect of a acute administration of EPO on insulin resistance and/or substrate metabolism in muscle tissue.

DETAILED DESCRIPTION:
Recently EPO receptors have been found in human muscle tissue, but what is still not known is what the physiological role of these receptors are. It has previously been shown that Growth Hormone mediate insulin resistance. The GH receptor and EPO receptor belong to the same family of cytokine receptors, and thereby share many of the same signalling pathways. In this study we want to investigate if there is a similar effect on insulin resistance and/or substrate metabolism after acute administration of EPO in human muscle tissue. Different signalling pathways are investigated på western blotting, and insulin sensitivity are measured be a hyperinsulinemic euglycemic clamp, and substrate metabolism is measured by the forearm model.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons
* Between 18 and 30 years
* Normal weight (BMI: 18-25)

Exclusion Criteria:

* Severe heart disease (NYHA 3)
* Uncontrolled hypertension
* Previous cerebrovascular disease
* Proliferative retinopathy
* Diabetes
* Musculo-skeletal diseases

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 4 and 6 hours post

SECONDARY OUTCOMES:
Substrate metabolism | 4 and 6 hours post

CONTACTS AND LOCATIONS:
Locations (1):
- Medicinsk forsknings laboratorium, Århus C, Denmark